CLINICAL TRIAL: NCT04092517
Title: MORINGA; Delivering Nutrition and Economic Value to the People of Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UAberdeen
Record Dates: First submitted 2018-10-15; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Malnourishment
Keywords: phytochemicals; systemic circulation
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Corn Soya Diet (Active Comparator): Control Corn Soya Diet will be prepared to a formulation for Corn Soya Blend (SUPER CEREAL) product adopted by the WFP as complementary food for children over than 6 months.
  Interventions: Other: Control Corn Soya Diet
- Test Corn Moringa Diet (Experimental): Test Corn Moringa Diet will be prepared to the same formulation as Corn Soya Blend, but the Soya content will be replaced with Moringa and no micronutrient premix will be added.
  Interventions: Other: Test Corn Moringa Diet

INTERVENTIONS:
Other: Control Corn Soya Diet — Ingredients (% by weight): Maize (78.30); Whole soya beans (20.00); Vitamin/Mineral FBF-V-13 (0.20); Dicalcium Phosphate anhydrous (1.23); Potassium chloride (0.27)
  Arms: Control Corn Soya Diet
Other: Test Corn Moringa Diet — Ingredients (% by weight): Maize (78.30); Moringa (20.0)
  Arms: Test Corn Moringa Diet

SUMMARY:
Lack of adequate nutrition is the single biggest contributor to child mortality. Malawi is amongst the countries most affected.

In global feeding programmes several variations of fortified blended foods are used and imported into the country of need as supplementary foods. However, the accessibility and efficacy of supplementary feeding is variable and can be a limiting factor for success in preventing and treating malnutrition. Therefore, in countries with widespread hunger, an increasing demand exists for innovative strategies offering alternative solutions for year-round access to commonly consumed home-grown products with good nutritional value.

Moringa Oleifera - described as 'a nutritional and medicinal cornucopia' is common throughout in Malawi. Moringa leaves can be repeatedly cropped and are rich source of nutrients and non-nutrient bioactive compounds. These nutritional characteristics give Moringa the potential to significantly contribute in Malawi's battle against malnutrition and mineral element deficiencies.

The aim of this study is to compare Moringa as a substitute in specially formulated supplementary foods in order to evaluate the in vivo bioavailability of key nutrients and bioactives and biological activities of the plant. This would assess the potential for establishing Moringa oleifera as an economically viable crop which could contribute towards establishing a resilient food supply chain in Malawi that will deliver essential nutrients across the population.

DETAILED DESCRIPTION:
Lack of adequate nutrition remains the world's most prevalent health problem and the single biggest contributor to child mortality. It is a direct or indirect cause of 43% deaths worldwide among children under 5 years of age. The two separate forms of malnutrition - wasting (a deficit in weight relative to length) and stunting (a deficit in length relative to age) are closely related and often occur together in the same children, leading to an increased risk of mortality. Although the prevalence of stunting is decreasing worldwide, Africa faces a rise in the absolute number of stunted children. Malawi is amongst the countries most affected in sub-Saharan Africa with 42% of the children being stunted and 4% wasted.

Maize is the principal food crop and dietary staple in many parts of the developing world including Malawi. This reliance on maize and the lack of dietary diversity is a significant contributing factor to micronutrient deficiencies (present in over 30 percent of the population).

Supplementary feeding by provision of extra nutrient-dense food beyond the home diet is an intervention aimed at improving the nutritional status or preventing the nutritional deterioration of the target population. Multiple socioeconomic and cultural factors play a role in determining the type and content of supplementary foods provided in different countries. The acceptability and efficacy of the nutrition support is variable (depending on sensory perception of the food, price, convenience of preparation, etc.) and can be a limiting factor for success in preventing and treating moderate and severe acute malnutrition. In this context there is an increasing demand for innovative strategies offering alternative solutions for year-round access to commonly consumed home-grown products with good nutritional value in countries with widespread hunger.

Moringa Oleifera - widely regarded as the 'miracle tree' has been described as 'a nutritional and medicinal cornucopia'. The Moringa plant is native to Northern India but has become naturalized in Malawi where it is common throughout. All parts of the plant are usable for different purposes, but for human and animal nutrition the leaves are the most widely utilised. Moringa leaves can be repeatedly and sustainably cropped and are rich in macro- and micronutrients, as well as bioactive compounds. These nutritional characteristics give Moringa the potential to significantly contribute in Malawi's battle against protein-energy malnutrition and mineral element deficiencies, providing home-grown feed and food products to replace/partly replace, with economic advantage, imported nutrient premixes.

Research devoted to nutritional characterisation of Moringa oleifera shows that it is a rich source of affordable, readily available, essential nutrients and phytoconstituents. The Moringa foliage is a good source of minerals, carotenoids and tocopherols, polyunsaturated fatty acids, ascorbic acid, folate and phenolics. Studies in animal models report significantly higher bioavailability for iron from Moringa foliage when compared to ferric citrate. Additionally, some major forms of folates were found to be highly bioavailable compared to other folate-rich foods, such as green leafy vegetables. However, different factors such as environmental, genetic, postharvest handling, stage of leaf development - significantly influence nutrient contents of Moringa leaves.

In human studies conducted with Moringa Oleifera to date, no adverse effects are reported and in many parts of the world its use as a food fortificant is on the increase. However, although many studies report improvement in the nutritional value of foods fortified with Moringa Oleifera, none of them show the digestibility (in-vivo or in-vitro) and nutrient bioavailability and high-quality research on its proposed nutritional and health benefits is currently scarce.

There are several variations (continuously refined to better meet the nutritional needs of beneficiaries) of currently endorsed fortified blended foods (FBF) used in global feeding programmes and imported into the country of need. Corn Soya Blend (CSB) fortified with a vitamin and mineral premix (SUPER CEREAL) is one such combination provided by the World Food Programme (WFP). The premix formula used may meet the minimum international standards, but is manufactured using inorganic compounds, which may not be fully bioavailable.

To the investigators' knowledge no human intervention trials have attempted to compare Moringa as modification substitute in specially formulated supplementary foods in order to evaluate in vivo bioavailability of key nutrients and bioactives and biological activities of the plant. This would give the potential for development for alternative formulations for locally produced supplementary foods.

Therefore, in this study the investigators aim to assess the nutritional composition of Moringa leaves (grown in three different sites in Malawi) in terms of macro-, micro- and non-nutrient composition. The sample with the most favourable profile will be used in a subsequent human intervention study. With this randomised, controlled, crossover-design study the investigators aim to evaluate the bioavailability potential of Moringa oleifera in terms of key nutrients and bioactives when compared with the current nutrient supplement SUPER CEREAL.

This human study is part of a wider collaborative study "MORINGA; delivering nutrition and economic value to the people of Malawi", investigating the possibility of establishing Moringa oleifera as an economically viable crop which will contribute towards launching a resilient food supply chain in Malawi that will deliver essential nutrients across the population.

Scientifically proven nutritive benefits of locally grown in Malawi Moringa oleifera could help to replace currently imported nutrients and products and develop sustainable production of a high-protein, micronutrient rich crop.

Two types of diets will be prepared:

Control meal: Corn Soya Blend Test meal: Corn Moringa Blend

In an acute intervention, these two test meals will allow us to evaluate the bioavailability of key nutrients and bioactives provided by Corn Moringa Blend when compared with Corn Soya Blend fortified with by an addition of a Micronutrient Premix.

In a cross-over fashion subjects will be randomly allocated to consume the Corn Moringa Blend or the Corn Soya/Micronutrient Premix Blend test meal. The volunteers will be invited to return to the Human Nutrition Unit (HNU) of the Rowett Institute for two intervention sessions. Both intervention sessions will be identical in all aspects except for the composition of the experimental meals.

For the duration of the intervention session (over 24 hour period), the volunteers will be asked to continue the low phytochemical diet and only consume water for the first five hours following consumption of the test meal. Each treatment session will be followed by at least one week wash-out period before crossing over to the second treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females;
* BMI 18-35;
* Age 18+

Exclusion Criteria:

* Subjects are taking prescribed medication;
* Subjects are pregnant or breastfeeding;
* Have given a blood donation in the last three months;
* Are unable to give written informed consent;
* Have eating disorders such as anorexia, bulimia, binge eating or night eating syndrome;
* Report any significant health issue;
* Subjects are taking vitamin or mineral supplements (unless they agree to discontinue supplementation 2wk before the start of the study);
* Food allergies/intolerances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in concentration of phytochemical metabolites in the systemic circulation | up to 24 hours
  Difference in concentration of phytochemical metabolites between baseline and postprandial states

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Russell, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No